CLINICAL TRIAL: NCT06854276
Title: A Randomized, Open-Label, Active-Controlled, Multicenter Phase II/III Clinical Study to Evaluate the Safety and Efficacy of SSS06 in the Treatment of Chemotherapy-Induced Anemia in Patients with Non-Myeloid Malignancies
Brief Title: Study of SSS06 for Chemotherapy-Induced Anemia in Non-Myeloid Malignancies
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSS06-202
Record Dates: First submitted 2025-02-11; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Chemotherapy-induced Anemia; Non-myeloid Malignancies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low-dose group (Experimental): SSS06, 200 μg, administered every 3 weeks, given 4 times
  Interventions: Drug: SSS06
- medium-dose group (Experimental): SSS06, 500 μg, administered every 3 weeks, given 4 times
  Interventions: Drug: SSS06
- high-dose group (Experimental): SSS06, 800 μg, administered every 3 weeks, given 4 times
  Interventions: Drug: SSS06
- Positive control group (Placebo Comparator): EPO, 36000 IU, administered every weeks, given 12 times
  Interventions: Drug: rhEPO

INTERVENTIONS:
Drug: SSS06 — SSS06 is a highly glycosylated, long-acting recombinant protein product produced through recombinant gene technology by introducing site-specific mutations into the rHuEPO gene.
  Arms: Low-dose group; high-dose group; medium-dose group
Drug: rhEPO — a recombinant human erythropoietin injection.
  Other Names: Yibiao
  Arms: Positive control group

SUMMARY:
This study employs a multicenter, randomized, open-label, positive drug-controlled, multiple ascending dose clinical trial design to comprehensively evaluate the safety, tolerability, immunogenicity, and pharmacokinetic characteristics of SSS06 injection in patients with chemotherapy-induced anemia from non-myeloid malignancies, while also exploring its potential efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥18 years at the time of signing the informed consent.
* Histologically or cytologically confirmed diagnosis of non-myeloid malignancies.
* Chemotherapy-induced anemia defined as hemoglobin (Hb) ≤100 g/L at screening, with a documented decrease in Hb of ≥10 g/L post chemotherapy initiation, as judged by the investigator.
* Serum ferritin ≥50 ng/mL and transferrin saturation (TSAT) ≥10% at screening.
* Body weight ≥40 kg at screening.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 1 or 2 at screening.
* Expected survival ≥6 months.
* Planned to receive at least 8 weeks of myelosuppressive chemotherapy starting from Day 1 of the study.
* Childbearing women must agree to use reliable contraception and have no plans to conceive or donate eggs from the start of study drug administration until 6 months post-last dose. Men must agree to use reliable contraception and have no plans to father a child or donate sperm from the start of study drug administration until 6 months post-last dose.
* Voluntarily sign informed consent, willing to participate in the trial, and able to comply with the protocol requirements for administration and follow-up, including examinations, visits, and other procedures.

Exclusion Criteria:

* Patients undergoing myelosuppressive chemotherapy with an expected curative outcome.
* Subjects receiving only hormone therapy, biologics, immunosuppressants (e.g., PD-1 and PD-L1 immune checkpoint inhibitors), or targeted therapies, or radiation therapy to treat/control their tumors; however, subjects receiving chemotherapy in combination with these therapies may be included.
* Subjects with a hematocrit (HCT) ≥ 36%.
* Subjects who have undergone interventions (e.g., blood transfusion, erythropoiesis-stimulating agents (ESAs), or hypoxia-inducible factor prolyl hydroxylase inhibitors (HIF-PHIs)) to elevate hemoglobin (Hb) levels to meet chemotherapy safety standards prior to the initiation of the scheduled chemotherapy regimen.
* Subjects who received red blood cell (RBC) transfusions, ESAs, or HIF-PHIs within 4 weeks prior to enrollment.
* Subjects with abnormal liver or kidney function test results: alanine aminotransferase (ALT) > 3×ULN, aspartate aminotransferase (AST) > 3×ULN, or total bilirubin (TBL) > 1.5×ULN (subjects with TBL up to 2×ULN may be included if ALT/AST are within normal limits and the investigator deems no safety concerns). Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m² (calculated using the CKD-EPI formula).
* Subjects with active systemic infections requiring treatment.
* Subjects with a history of clinically significant cardiovascular disease, including New York Heart Association (NYHA) Class III or IV heart failure within the past 6 months, uncontrolled hypertension or hypotension, or severe valvular or endocardial disease history that may increase the risk of thromboembolic events.
* Subjects who experienced thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism, myocardial infarction, stroke, transient ischemic attack) within the past 6 months.
* Subjects with clinically significant anemia due to other causes, such as iron deficiency, vitamin B12 or folate deficiency, autoimmune anemia, hemolysis, hemorrhage, or genetic anemias (e.g., sickle cell anemia or thalassemia).
* Subjects with clinically significant or uncontrolled chronic inflammatory or autoimmune diseases (e.g., rheumatoid arthritis, Crohn's disease, celiac disease).
* Subjects with severe or active liver disease.
* Subjects planning to undergo major surgery during the treatment period (surgery with minimal blood loss that does not affect Hb concentration is exempt).
* Subjects with myeloid malignancies.
* Subjects with primary or metastatic malignant tumors in the central nervous system.
* Subjects testing positive for human immunodeficiency virus (HIV) antibodies or syphilis antibodies.
* Subjects positive for hepatitis B virus (HBV) or hepatitis C virus (HCV):

  1. Subjects with inactive HBsAg carriers or stable hepatitis B patients (HBV DNA < 500 IU/mL) may be included, with regular monitoring of HBV DNA during the study as recommended by the investigator.
  2. Subjects with HCV antibody positivity (HCV-Ab+) may be included if HCV RNA is negative, with regular monitoring of HCV RNA during the study as recommended by the investigator.
* Subjects who have used any investigational drugs within 4 weeks prior to Day 1 of treatment or plan to use such drugs during the clinical trial.
* Subjects with a history of alcoholism, drug abuse, or addiction.
* Subjects deemed unsuitable for participation in the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) Events (NCI-CTCAE V5.0). | From Day 1 to Day 113
  All adverse events occurring during the entire study period will be assessed and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE Version 5.0).

SECONDARY OUTCOMES:
Concentration of hemoglobin maximum change from baseline | From Day 1 to Day 113
  the maximum change in Hb from baseline within 13 weeks without red blood cell transfusion.

IPD SHARING:
Plan to Share IPD: No